CLINICAL TRIAL: NCT00563576
Title: Pilot Study of Femring Estrogen Supplementation During Depo-Provera Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAC6363
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Metrorrhagia
Keywords: Depo-Provera; Medroxyprogesterone Acetate; Metrorrhagia; Irregular Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Estradiol; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Depo-Provera/Femring (Experimental): Subjects will receive an estrogen vaginal ring (100 mcg) during the first 90 days of Depo-Provera use.
  Interventions: Drug: Femring®; Drug: DepoProvera ®
- Depo-Provera Injection Alone (Other): Subjects will receive Depo-Provera intramuscular injection.
  Interventions: Drug: DepoProvera ®

INTERVENTIONS:
Drug: Femring® — Estrogen vaginal ring (100 mcg) placed for the first 90 days of Depo-Provera use.
  Femring® (estradiol acetate vaginal ring) is a flexible off-white ring designed for vaginal insertion with measurements that include an outer diameter of 56 mm, cross-sectional diameter of 7.6 mm, and core diameter of 2 mm. Femring® 0.1 mg/day has a central core containing 24.8 mg of estradiol acetate which releases at a rate equivalent to 0.1 mg of estradiol per day for 3 months.
  Other Names: Estradiol Acetate Vaginal Ring
  Arms: Depo-Provera/Femring
Drug: DepoProvera ® — Medroxyprogesterone intramuscular injection comes as a suspension (liquid) to be injected into the buttocks or upper arm. It is usually given once every 3 months (13 weeks), and the recommended dose is 150 mg.
  Other Names: Depot Medroxyprogesterone Acetate (DMPA)

SUMMARY:
Many women choose Depo-Provera for birth control because it is easy to use and very effective. However, a significant number of Depo-Provera users experience irregular bleeding during the first 90 days. Many users discontinue after their first injection due to irregular bleeding. This study will evaluate the effect of using an estrogen vaginal ring during the first 90 days of Depo-Provera use to see if it is acceptable to women and whether it decreases irregular bleeding during the first 90 days of use and increases continuation to a second injection.

DETAILED DESCRIPTION:
Many women choose depot medroxyprogesterone acetate (DMPA) for contraception because it is long-acting, highly effective, and requires minimal user involvement. One of the most common side effects of DMPA use during the first 90 day cycle is irregular bleeding. There are few studies that report mean number of bleeding days among DMPA users. A large World Health Organization (WHO) trial including ten international centers and menstrual data on 748 women using DMPA including 372 woman-years of follow-up reported 23.6 mean days of spotting and bleeding during the first cycle with a standard deviation of 18.9 days (WHO). Another study sponsored by WHO (n=575) reported that 25% of subjects had bleeding/spotting episodes during the first cycle of DMPA that exceeded 13 days. The number of bleeding/spotting days and number of bleeding/spotting episodes decreased over successive reference periods (Said 1987).

Discontinuation rates are high after the first injection and related to irregular bleeding. Rates of discontinuation after the first injection range from 15-60% but were around 30% in most studies (Harel, Paul, Polaneczy, Lim, Hubacher, Sangi, Rickert). Several studies noted that the largest percentage of discontinuation during the first year of DMPA use occurs after the first injection (Rickert, Hubacher, Lim). Irregular bleeding is uniformly cited as one of the most common reasons for discontinuation, accounting for 17-60% of all reasons given (Harel, Paul, Polaneczy, Lim, Sangi). An intervention to prevent or minimize irregular bleeding during the first 90 days of DMPA use could potentially minimize or prevent this bothersome side effect and thus improve continuation.

Few studies have examined the effect of prophylactic or therapeutic estrogen supplementation on irregular bleeding in DMPA users. A randomized trial (n=132) of cyclic transdermal estradiol 0.1 mg/day (Climara) for 3 months versus placebo in women initiating DMPA immediately post-abortion showed no difference in continuation rates at 12 months; however, the authors of this study reported a high rate of non-compliance with the study protocol and lacked an adequate sample size to detect a difference (Goldberg). This is the only study to report on prophylactic estrogen supplementation in DMPA users.

Two studies evaluated therapeutic estrogen supplementation in DMPA users. In 1996, WHO published results of a trial in which women using DMPA and experiencing a bleeding episode greater than 7 days during the first or second injection interval were offered treatment. Subjects (n=278) were randomized to a 14 day course of 50 mcg ethinyl estradiol, 2.5 mg oestrone sulphate, or placebo. The authors found that subjects treated with ethinyl estradiol had shorter median time to cessation of bleeding and fewer bleeding/spotting days (Said 1996). An observational study (n=131) of adolescents reporting vaginal bleeding on DMPA who were treated with monophasic oral contraceptive pills identified improvement of bleeding patterns and a high rate of continuation in those receiving treatment (Rager).

Estrogen supplementation appears to be more effective than placebo in stopping and decreasing bleeding in Norplant users. Women who presented with a spontaneous complaint of prolonged or irregular bleeding were randomly assigned to receive 20 days of treatment with a combined oral contraceptive, 50 mcg ethinyl estradiol, or placebo. Both combined oral contraceptive pills and estradiol were significantly more effective than placebo in stopping bleeding and decreasing the mean number of bleeding days during treatment (Alvarez).

To summarize, prior studies have not identified an acceptable or effective prophylactic intervention to prevent or minimize irregular bleeding or improve continuation rates in DMPA users. The first cycle of DMPA is a critical time for such an intervention. Our study will evaluate estrogen supplementation with an estrogen vaginal ring during the first 90 days of DMPA use versus no estrogen supplementation and report on acceptability, bleeding patterns, and continuation rates. Femring®, an estradiol vaginal ring currently used for treatment of postmenopausal symptoms, provides 100 mcg of estradiol per day with one ring designed for 90 days of consecutive use. This dose provides systemic levels sufficient to suppress vasomotor symptoms in postmenopausal women (Speroff). The vaginal ring would require minimal user involvement when placed at the time of DMPA initiation. If acceptable and effective, this intervention could prevent or minimize irregular bleeding and improve continuation rates of this highly effective contraceptive method.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older who are initiating Depo-Provera for contraception
* English or Spanish-speaking
* Have a negative urine pregnancy test

Exclusion Criteria:

* Contraindications to either Depo-Provera or Femring (estrogen vaginal ring)
* Have used Depo-Provera or Mirena in the prior 6 months
* Have had an induced abortion, spontaneous abortion, or birth in prior 8 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Dempsey, MD, MPH, Principal Investigator — Medical University of South Carolina; Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Title X Family Planning Clinic, New York, New York, United States

REFERENCES:
- [Background] Alvarez-Sanchez F, Brache V, Thevenin F, Cochon L, Faundes A. Hormonal treatment for bleeding irregularities in Norplant implant users. Am J Obstet Gynecol. 1996 Mar;174(3):919-22. doi: 10.1016/s0002-9378(96)70326-5. PMID 8633669
- [Background] Belsey EM, Machin D, d'Arcangues C. The analysis of vaginal bleeding patterns induced by fertility regulating methods. World Health Organization Special Programme of Research, Development and Research Training in Human Reproduction. Contraception. 1986 Sep;34(3):253-60. doi: 10.1016/0010-7824(86)90006-5. PMID 3539509
- [Background] Dieben TO, Roumen FJ, Apter D. Efficacy, cycle control, and user acceptability of a novel combined contraceptive vaginal ring. Obstet Gynecol. 2002 Sep;100(3):585-93. doi: 10.1016/s0029-7844(02)02124-5. PMID 12220783
- [Background] Goldberg AB, Cardenas LH, Hubbard AE, Darney PD. Post-abortion depot medroxyprogesterone acetate continuation rates: a randomized trial of cyclic estradiol. Contraception. 2002 Oct;66(4):215-20. doi: 10.1016/s0010-7824(02)00391-8. PMID 12413614
- [Background] Harel Z, Biro FM, Kollar LM, Rauh JL. Adolescents' reasons for and experience after discontinuation of the long-acting contraceptives Depo-Provera and Norplant. J Adolesc Health. 1996 Aug;19(2):118-23. doi: 10.1016/1054-139X(95)00322-J. PMID 8863083
- [Background] Hubacher D, Goco N, Gonzalez B, Taylor D. Factors affecting continuation rates of DMPA. Contraception. 1999 Dec;60(6):345-51. doi: 10.1016/s0010-7824(99)00104-3. PMID 10715369
- [Background] Lim SW, Rieder J, Coupey SM, Bijur PE. Depot medroxyprogesterone acetate use in inner-city, minority adolescents: continuation rates and characteristics of long-term users. Arch Pediatr Adolesc Med. 1999 Oct;153(10):1068-72. doi: 10.1001/archpedi.153.10.1068. PMID 10520615
- [Background] Novak A, de la Loge C, Abetz L, van der Meulen EA. The combined contraceptive vaginal ring, NuvaRing: an international study of user acceptability. Contraception. 2003 Mar;67(3):187-94. doi: 10.1016/s0010-7824(02)00514-0. PMID 12618252
- [Background] Paul C, Skegg DC, Williams S. Depot medroxyprogesterone acetate. Patterns of use and reasons for discontinuation. Contraception. 1997 Oct;56(4):209-14. doi: 10.1016/s0010-7824(97)00140-6. PMID 9408701
- [Background] Polaneczky M, Liblanc M. Long-term depot medroxyprogesterone acetate (Depo-Provera) use in inner-city adolescents. J Adolesc Health. 1998 Aug;23(2):81-8. doi: 10.1016/s1054-139x(98)00014-7. PMID 9714170
- [Background] Rager KM, Fowler A, Omar HA. Successful treatment of depot medroxyprogesterone acetate-related vaginal bleeding improves continuation rates in adolescents. ScientificWorldJournal. 2006 Mar 19;6:353-5. doi: 10.1100/tsw.2006.69. PMID 16547584
- [Background] Rickert VI, Tiezzi L, Lipshutz J, Leon J, Vaughan RD, Westhoff C. Depo Now: preventing unintended pregnancies among adolescents and young adults. J Adolesc Health. 2007 Jan;40(1):22-8. doi: 10.1016/j.jadohealth.2006.10.018. PMID 17185202
- [Background] Said S, Omar K, Koetsawang S, Kiriwat O, Srisatayapan Y, Kazi A, Ajmal F, Wynter HH, Pretnar-Darovec A, Benitez IB. A multicentered phase III comparative clinical trial of depot-medroxyprogesterone acetate given three-monthly at doses of 100 mg or 150 mg: II. The comparison of bleeding patterns. World Health Organization. Task Force on Long-Acting Systemic Agents for Fertility Regulation Special Programme of Research, Development and Research Training in Human Reproduction. Contraception. 1987 Jun;35(6):591-610. doi: 10.1016/s0010-7824(87)80019-7. PMID 2959448
- [Background] Said S, Sadek W, Rocca M, Koetsawang S, Kirwat O, Piya-Anant M, Dusitsin N, Sethavanich S, Affandi B, Hadisaputra W, Kazi A, Ramos RM, d'Arcangues C, Belsey EM, Noonan E, Olayinka I, Pinol A. Clinical evaluation of the therapeutic effectiveness of ethinyl oestradiol and oestrone sulphate on prolonged bleeding in women using depot medroxyprogesterone acetate for contraception. World Health Organization, Special Programme of Research, Development and Research Training in Human Reproduction, Task Force on Long-acting Systemic Agents for Fertility Regulation. Hum Reprod. 1996 Oct;11 Suppl 2:1-13. doi: 10.1093/humrep/11.suppl_2.1. PMID 8982739
- [Background] Sangi-Haghpeykar H, Poindexter AN 3rd, Bateman L, Ditmore JR. Experiences of injectable contraceptive users in an urban setting. Obstet Gynecol. 1996 Aug;88(2):227-33. doi: 10.1016/0029-7844(96)00194-9. PMID 8692507
- [Background] Speroff L. Efficacy and tolerability of a novel estradiol vaginal ring for relief of menopausal symptoms. Obstet Gynecol. 2003 Oct;102(4):823-34. doi: 10.1016/s0029-7844(03)00764-6. PMID 14551014
- [Background] Multinational comparative clinical evaluation of two long-acting injectable contraceptive steroids: noresthisterone oenanthate and medroxyprogesterone acetate. 2. Bleeding patterns and side effects. Contraception. 1978 May;17(5):395-406. PMID 657807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a Title X Family Planning Clinic in New York City.
Pre-assignment Details: Women seeking DMPA eligible to participate it 18 years old, English or Spanish speaking, had not used DMPA or Levonorgestrel intrauterine system in the preceeding 120 days. Women reporting oligomenorrheas (defined as fewer that 4 periods in the last 6 months), amenorrhea, or contraindications to either DMPA or estrogen were excluded.
Groups:
- Femring: Subjects will receive an estrogen vaginal ring (100mcg) during the first 90 days of Depo-Provera use.
- Depot Medroxyprogesterone Acetate (DMPA) Alone: Subjects will receive Depo-Provera intramuscular injection.
Period: Overall Study
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Started | 35 | 36
Completed | 21 | 22
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Bleeding or Spotting Days
Description: Bleeding and spotting were defined using World Health Organization criteria and measured through daily diaries given to participants and collected at the 3 and 6 month followup. In addition, a study staff member called participants weekly to collect the daily bleeding and spotting calendar for that week to optimize the accuracy of this information.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Number analyzed (Participants) | 35 | 36
days | 16 (0.19) | 28 (0.19)

2. Secondary Outcome: Percentage of Users Who Were Satisfied With Femring
Description: Acceptability was measured using questionnaires that assessed satisfaction of Femring and usage of the ring. This outcome was only measured among the intervention group of women who actually were randomized to use of Femring. Acceptability of the vaginal ring was high among those in the intervention group.
Time Frame: 3 months
Population: Acceptability was reported among the 26 participants in the Femring group who were available for followup, i.e., per protocol.
Measure: Number; unit: participants
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Number analyzed (Participants) | 26 | 0
participants | 84 |

3. Secondary Outcome: Number of Subjects Who Receive a 2nd Injection of Depo-Provera
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Number analyzed (Participants) | 35 | 36
participants | 20 | 16

4. Secondary Outcome: Percentage of Subjects Who Receive a 3rd Injection
Time Frame: 6 months
Population: Only the women who completed the study up to the secondary endpoint were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Number analyzed (Participants) | 17 | 16
Participants | 13 | 10

ADVERSE EVENTS:
Arm/Group | Femring | Depot Medroxyprogesterone Acetate (DMPA) Alone
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No